CLINICAL TRIAL: NCT07320755
Title: Analysis of Computed Tomography Derived Maps for Determining Changes of the Liver Volume After Exposure to Radiotherapy
Acronym: ACT-LIVERT
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alzahraa Ahmed Fouad, Principal Investigator, Assiut University
Other Study IDs: RAD-LIVER-2025
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Intra-abdominal Malignancies; Liver as Organ at Risk; Radiation-related Liver Changes
Keywords: liver volume changes after radiotherapy; CT-derived volumetric analysis; Hepatic toxicity prediction; Radiotherapy planning optimization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Radiotherapy is commonly used to treat cancers involving the liver or nearby organs. While effective, radiation exposure can affect healthy liver tissue and may lead to changes in liver size and function. Monitoring these changes is important to improve treatment planning and reduce the risk of liver-related complications.

This study aims to evaluate changes in liver volume using computed tomography (CT) imaging before and after radiotherapy. By analyzing CT-derived liver maps, the study seeks to better understand how the liver responds to radiation treatment over time.

The study will include patients who undergo radiotherapy and have CT imaging performed as part of their routine clinical care. No additional procedures or treatments will be required for participation. The findings of this study may help improve future radiotherapy planning and patient monitoring by providing better information on liver volume changes following radiation exposure.

DETAILED DESCRIPTION:
Radiotherapy plays a central role in the management of primary and metastatic tumors involving the liver or adjacent anatomical regions. Despite advances in radiation delivery techniques, the liver remains a radiosensitive organ, and radiation-induced liver injury continues to be a clinically significant concern. Quantitative assessment of liver volume changes may provide valuable insight into hepatic response and tolerance to radiation exposure.

This study is designed to analyze computed tomography (CT)-derived liver volume maps to assess changes in liver volume following radiotherapy. CT images acquired as part of standard clinical practice will be used to generate volumetric measurements of the liver at baseline and during post-treatment follow-up. Advanced image analysis techniques will be applied to evaluate spatial and global liver volume changes.

The study is observational in nature and does not involve any investigational drugs or devices. All imaging data will be obtained from routine clinical workflows without modification to standard patient care. Demographic, clinical, and treatment-related parameters may be correlated with observed liver volume changes to explore potential associations.

The results of this study are expected to enhance understanding of radiation-related hepatic effects and support optimization of radiotherapy planning strategies. Improved knowledge of liver volume dynamics may contribute to better prediction of treatment-related toxicity and support individualized patient management in future clinical practice.

ELIGIBILITY:
1. Inclusion criteria:

   * Adults aged 18 years or older.
   * Received radiation therapy (RT) involving the liver (e.g., SBRT, IMRT). The study involves patients in whom the liver was exposed to radiotherapy, either as a direct target (in hepatic-directed treatments as in HCC or liver metastasis) or indirectly as an organ-at-risk (OAR) during irradiation of nearby anatomical regions (as lower lung, gastric, or abdominal sites) where the liver was partially included within the radiation field.

   The analysis aims to evaluate radiation-induced volumetric changes regardless of whether the liver was the primary target or secondarily affected.
   * Availability of paired pre- and post-RT CT scans of sufficient quality.
   * 3D dose distribution data from the RT treatment plan.
   * Clinical follow-up data, including liver function tests and toxicity records.
   * No evidence of major anatomical changes between scans unrelated to RT (e.g., surgery).
2. Exclusion criteria:

   * Patients with a history of major liver surgery (e.g., resection or transplant) between the pre- and post-RT scans.
   * Presence of severe motion artifacts or poor-quality CT scans that hinder accurate image analysis.
   * Incomplete or missing 3D radiation dose distribution data.
   * Lack of sufficient clinical follow-up information (e.g., liver function tests, toxicity outcomes).
   * Concurrent systemic therapies (e.g., chemotherapy or immunotherapy) during the imaging interval that may confound liver volume changes, unless controlled for in analysis.
   * Pre-existing liver conditions that could independently alter liver volume (e.g., cirrhosis, advanced hepatic steatosis) if not accounted for.
   * Patients under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who have received radiotherapy for liver or nearby tumors and have available pre-treatment and post-treatment CT imaging for assessment of liver volume changes. Both males and females are included, with a minimum age of 18 years and no upper age limit. Participants are selected based on availability of imaging data from routine clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Liver Volume After Radiotherapy | Liver volume changes will be assessed at post-treatment intervals, typically at 1, 3, and 6 months after radiotherapy. If only a single post-treatment scan is available, evaluation will occur approximately 3 months after treatment completion.
  The primary outcome is the quantitative change in liver volume measured using computed tomography (CT) imaging before and after radiotherapy. Liver volume will be assessed using standard imaging software and protocols, and changes will be calculated relative to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Amr Farouk Mourad, Prof., Study Chair — Assiut University; Omar Mostafa Mahmoud Mohammad, Assist Prof., Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study uses retrospective clinical imaging and patient records, and the data contain sensitive health information. Sharing is restricted to protect patient privacy and comply with institutional and ethical regulations.

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/40660871/